CLINICAL TRIAL: NCT02040623
Title: Phase 2, Multi-Center, Randomized, Double-Masked, Placebo-Controlled Clinical Study to Assess the Safety and Efficacy of 0.2% and 0.5% R932348 Ophthalmic Solutions for the Treatment of Keratoconjunctivitis Sicca in Patients With Chronic Ocular Graft Versus Host Disease
Brief Title: Safety and Efficacy Study of R932348 Ophthalmic Solution in Chronic Ocular Graft Versus Host Disease Patients(DROPS-2)
Acronym: DROPS-2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rigel Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C-932348-004
Record Dates: First submitted 2014-01-16; First posted 2014-01-20 (Estimated); Results first posted 2016-10-10 (Estimated); Last update posted 2016-10-10 (Estimated); Status verified 2016-08

CONDITIONS: Chronic Graft-versus-host Disease
Keywords: Chronic Graft versus Host Disease; Keratoconjunctivitis Sicca
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome; Keratoconjunctivitis Sicca

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- R348 Ophthalmic Solution, 0.2% (Active Comparator): R348 Ophthalmic Solution 0.2% 2 drops per eye twice a day
  Interventions: Drug: R348 Ophthalmic Solution, 0.2%
- R348 Ophthalmic Solution, 0.5% (Active Comparator): R348 Ophthalmic Solution, 0.5% 2 drops per eye twice a day
  Interventions: Drug: R348 Ophthalmic Solution, 0.5%
- Placebo (Placebo Comparator): Placebo Ophthalmic Solution 2 drops per eye twice a day
  Interventions: Other: Placebo Ophthalmic Solution

INTERVENTIONS:
Drug: R348 Ophthalmic Solution, 0.2% — R348 Ophthalmic Solution 0.2% 2 drops per eye twice a day
  Other Names: R932348
  Arms: R348 Ophthalmic Solution, 0.2%
Drug: R348 Ophthalmic Solution, 0.5% — R348 Ophthalmic Solution, 0.5% 2 drops per eye twice a day
  Other Names: R932348
  Arms: R348 Ophthalmic Solution, 0.5%
Other: Placebo Ophthalmic Solution — Placebo Ophthalmic Solution 2 drops per eye twice a day
  Arms: Placebo

SUMMARY:
* To assess the efficacy of R348 Ophthalmic Solutions administered for 12 weeks to subjects evaluated by objective and subjective measures.
* To investigate the safety and tolerability of R348 Ophthalmic Solutions administered for 12 weeks to subjects.

ELIGIBILITY:
Inclusion Criteria:

* Received an Allogeneic hematologic stem cell transplantation at least 3 months prior.
* Subjects with post Allogeneic hematologic stem cell transplantation onset or worsening of dry eye symptoms for at least 1 month prior.
* Use of over-the-counter and/or prescription eye drops for dry eye symptoms within 1 month.
* Corneal fluorescein staining score of ≥ 2 in 1 region and ≥ 1 in at least 1 other region.
* Total lissamine green conjunctival staining score (according to a modified National Eye Institute grading system) of ≥ 2.

Exclusion Criteria:

* Clinically unstable Graft versus Host Disease (requiring a change in immunosuppressive regimen), medical condition, or laboratory abnormality
* Used topical ophthalmic cyclosporine within 45 days.
* Used any topical ophthalmic steroid within 2 weeks.
* Used autologous serum eye drops within 2 weeks.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2014-03; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rigel Pharmaceuticals, Inc., Study Director — Rigel Pharmaceuticals,Inc.
Locations (2):
- United States (2):
  - U. Miami - Bascom Palmer Eye Institute, Plantation, Florida
  - Massachusetts Eye and Ear Infirmary, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | R348 Ophthalmic Solution, 0.2% | R348 Ophthalmic Solution, 0.5% | Placebo
Started | 11 | 12 | 12
Completed | 7 | 6 | 10
Not Completed | 4 | 6 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | R348 Ophthalmic Solution, 0.2% | R348 Ophthalmic Solution, 0.5% | Placebo | Total
Number analyzed (Participants) | 11 | 12 | 12 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.1 (9.34) | 55.8 (17.15) | 52.5 (15.96) | 55.13 (10.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 6 | 16
  Male | 6 | 7 | 6 | 19

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline (Visit 1) of Total Corneal Fluorescein Staining Score at 12 Weeks.
Description: Change from baseline (Visit 1) of total CFS score at 12 weeks. Total CFS score range 0-20, where '0' represents no fluorescein staining of any region and '20' represents severe staining the entire cornea.
Time Frame: Baseline to 12 weeks
Population: The per-protocol (PP) population excludes subjects with significant protocol deviations or with early study termination
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | R348 Ophthalmic Solution, 0.2% | R348 Ophthalmic Solution, 0.5% | Placebo
Number analyzed (Participants) | 7 | 6 | 9
units on a scale | -4.2 (2.9) | -6.2 (3.7) | -2.1 (2.6)

ADVERSE EVENTS:
Time Frame: The AE reporting period begins with the first dose of study drug and ends with the final study follow-up visit (Day 91).
Arm/Group | R348 Ophthalmic Solution, 0.2% | R348 Ophthalmic Solution, 0.5% | Placebo
Serious Adverse Events (participants affected / at risk) | 1/11 | 2/12 | 1/12
Other Adverse Events (participants affected / at risk) | 11/11 | 10/12 | 9/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | R348 Ophthalmic Solution, 0.2% (N=11) | R348 Ophthalmic Solution, 0.5% (N=12) | Placebo (N=12)
Hyperbilirubinaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Clostridium Difficile infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary Fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Microembolism (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | R348 Ophthalmic Solution, 0.2% (N=11) | R348 Ophthalmic Solution, 0.5% (N=12) | Placebo (N=12)
Hyperbilirubinaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Ocular Hyperaemia (Eye disorders) | 2 (4) | 0 (0) | 0 (0)
Blepharitis (Eye disorders) | 1 (1) | 1 (2) | 0 (0)
Corneal Deposits (Eye disorders) | 1 (2) | 0 (0) | 0 (0)
Dry Eye (Eye disorders) | 1 (2) | 0 (0) | 1 (2)
Eye Irritation (Eye disorders) | 1 (2) | 1 (2) | 1 (2)
Foreign Body Sensation in Eyes (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Posterior Capsule Opacification (Eye disorders) | 1 (2) | 0 (0) | 0 (0)
Punctate Keratitis (Eye disorders) | 1 (1) | 2 (3) | 2 (2)
Trichiasis (Eye disorders) | 1 (2) | 0 (0) | 1 (2)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 1 (2)
Cataract Nuclear (Eye disorders) | 0 (0) | 0 (0) | 1 (2)
Conjunctival Haemorrhage (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Conjunctival Hyperaemia (Eye disorders) | 0 (0) | 1 (1) | 1 (2)
Conjunctivitis (Eye disorders) | 0 (0) | 0 (0) | 1 (2)
Corneal Opacity (Eye disorders) | 0 (0) | 0 (0) | 1 (2)
Diplopia (Eye disorders) | 0 (0) | 1 (2) | 0 (0)
Eye Pain (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Eyelid Ptosis (Eye disorders) | 0 (0) | 0 (0) | 1 (2)
Iris Adhesions (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Keratitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Meibomian Gland Dysfunction (Eye disorders) | 0 (0) | 1 (1) | 1 (2)
Optic Nerve Cupping (Eye disorders) | 0 (0) | 0 (0) | 1 (2)
Retinal Pigmentation (Eye disorders) | 0 (0) | 0 (0) | 1 (2)
Vision Blurred (Eye disorders) | 0 (0) | 1 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (3) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomitting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Instillation Site Pain (General disorders) | 2 (4) | 0 (0) | 0 (0)
Instillation Site Foreign Body Sensation (General disorders) | 0 (0) | 1 (2) | 0 (0)
Secretion Discharge (General disorders) | 0 (0) | 1 (2) | 0 (0)
Cholangitis Sclerosing (Hepatobiliary disorders) | 1 (2) | 0 (0) | 0 (0)
Seasonal Allergy (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Graft Versus Host Disease (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
Arthritis Bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Oral Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Skin Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Clostridium Difficile Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Dacryocystitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 3 (3) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Arthropod Bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Intraocular Pressure Increased (Investigations) | 1 (2) | 0 (0) | 0 (0)
Blood Triglycerides Increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Diabetes Mellitus (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Restlessness (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Acute Kidney Injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Parosmia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary Fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory Tract Irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Microembolism (Vascular disorders) | 1 (1) | 1 (1) | 1 (1)
Ecchymosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperaemia (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No